CLINICAL TRIAL: NCT01961739
Title: Double Blinded Randomized Clinical Trial of the Efficacy of Topical 2% Lidocaine for the Treatment of Symptomatic Hemorrhoids
Brief Title: Topical 2% Lidocaine for the Treatment of Symptomatic Hemorrhoids
Acronym: H1-5
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Dubrava (Other)
Collaborators: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Principal Investigator, Mario Kopljar, Dr. sc., University Hospital Dubrava
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PROTOCOL H1-5
Record Dates: First submitted 2013-10-09; First posted 2013-10-11 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Hemorrhoids
Keywords: Hemorrhoids; Lidocaine
MeSH Terms: conditions — Hemorrhoids | interventions — Lidocaine; Petrolatum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2% lidocaine (Experimental): topical application, two times per day for 15 consecutive days
  Interventions: Drug: 2% lidocaine
- placebo (Placebo Comparator): vaseline base applied topically, two times per day for 15 consecutive days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: 2% lidocaine — Topical application, twice per day for 15 consecutive days
  Other Names: lidocaine
  Arms: 2% lidocaine
Drug: placebo — topical application, twice per day for 15 consecutive days
  Other Names: vaseline
  Arms: placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of topical 2% lidocaine in the therapy of symptomatic hemorrhoids. Efficacy will be determined by:

1. the change from baseline in pain, itching, bleeding, swelling, discomfort, general well-being and improvement since the beginning of treatment as separate components of CORRECTS scale
2. the change in overall CORRECTS values from baseline
3. the change in degree of hemorrhoids from baseline

DETAILED DESCRIPTION:
This is a double blinded randomized clinical study into the effect of topical 2% lidocaine in patients with symptomatic hemorrhoids.

Calculated sample size is 69 patients per arm, based on expected improvement of pain and healing by 30% at p<0.05 and power goal of 95%. Taking into account a drop-out rate of 50%, total number of 69 patients in each arm is estimated as sufficient to close the study.

Patients will be randomly assigned into 2 arms, arm 1 (treatment): topical 2% lidocaine and arm 2 (control): vaseline base. Each arm will consist of 69 patients. Patients will be assigned to either treatment or control arm according to the randomization table.

* Treatment arm - topical 2% lidocaine. Topical application of 2% lidocaine in vaseline base repeated two times per day,
* Control arm - vaseline base. Topical application of pure vaseline base twice per day.

In addition to the aforementioned topical treatments, all patients will be given written instructions to perform dietary modifications and anal hygiene. All patients with bleeding hemorrhoids will be given Detralex 2 tablets twice per day.

Those patients in whom a technically successful procedure has been completed will be considered as valuable for the efficacy evaluation. A technically successful procedure is defined as the completion of treatment procedures stipulated in this protocol and consists of correct drug dose and frequency of application, adherence to written instructions for dietary modification and anal hygiene and presence at follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* clinically present enlarged hemorrhoids, grade 1-4 (for definition see Appendix 1)
* symptoms of pain or itching
* age 18 years or more
* willing and able to comply with the study
* geographically suitable, meaning with reliable transportation for outpatients to the testing site

Exclusion Criteria:

* actual pregnancy
* inability to provide informed consent
* any anal topical medication applied in the last 7 days
* any anal surgery (including surgical or instrumental procedures defined in the section 4.3) in the last 60 days
* known allergy to vaseline, lidocaine or Dulcolax
* other anal disorders and diseases including Crohns disease, ulcerative colitis, undefined inflammatory bowel disease, anal fissures, perianal fistulas, perianal rash or eczema, rectal prolapse, rectocele, benign or malignant anal and rectal tumor and perianal infections
* contraindication for topical anal application of vaseline or lidocaine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Change in CORRECTS scale | 15 days after treatment initiantion
  Change in CORRECTS scale and grade of haemorrhoids

SECONDARY OUTCOMES:
Percentage of adverse events | within 15 days after treatment initiation
  Secondary objective is to assess the safety and tolerability of [TREATMENT] by determining:
  1. percentage of adverse events (complications)
  2. percentage of treatment discontinuations due to adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Mario Kopljar, MD, PhD, Principal Investigator — University Hospital Dubrava; Tihomir Kekez, Principal Investigator — Clinical Hospital Centre Zagreb
Locations (2):
- Croatia (2):
  - Clinical Hospital Centre Zagreb, Zagreb
  - Clinical Hospital Dubrava, Zagreb